CLINICAL TRIAL: NCT02234310
Title: An Open-Label, Multicenter Evaluation of the Safety and Efficacy of Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc; BIIB029) in the Prevention and Treatment of Bleeding in Previously Untreated Patients With Severe Hemophilia B
Brief Title: Study to Determine the Safety and Efficacy of rFIXFc in Previously Untreated Males With Severe Hemophilia B
Acronym: PUPs B-LONG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 998HB303; 2013-003629-27 (EudraCT Number)
Record Dates: First submitted 2014-07-17; First posted 2014-09-09 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia B
Keywords: prophylaxis treatment; episodic treatment
MeSH Terms: conditions — Hemophilia B | interventions — factor IX Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc) (Experimental): Participants received rFIXFc intravenous (IV) injection as follows: Prophylactic treatment regimen: started with rFIXFc 50 International Units per kilogram (IU/kg) weekly until a participant reached at least 50 exposure days (ED=24-hour period in which greater than or equal to (>=1) injection/dose of rFIXFc was given) to rFIXFc, withdrawal from study or end of study. Adjustments to dose and dosing interval was based on incremental recovery, subsequent Factor IX (FIX) levels, physical activity, bleeding pattern, in accordance with local standards of care for prophylactic regimen (PR). Treatment with episodic (on demand) regimen can be initiated before PR at investigators discretion. Episodic (On demand; optional): rFIXFc at individual doses based on participant's clinical condition, type and severity of bleeding event until PR.
  Interventions: Biological: rFIXFc

INTERVENTIONS:
Biological: rFIXFc — Adjustments to the dose and interval of rFIXFc was made in this study based on investigator discretion using available pharmacokinetic (PK) data, subsequent FIX trough and peak levels, level of physical activity, and bleeding pattern, in accordance with local standards of care for a prophylactic regimen. There was an option to start study dosing as episodic treatment (on-demand).
  Other Names: BIIB029; Alprolix; recombinant coagulation factor IX Fc fusion protein

SUMMARY:
The primary objective of the study was to evaluate the safety of recombinant coagulation factor IX Fc fusion protein (rFIXFc, BIIB029) in previously untreated patients (PUPs) with severe hemophilia B. Secondary objectives were to evaluate the efficacy of rFIXFc in the prevention and treatment of bleeding episodes in PUPs, and to evaluate rFIXFc consumption for prevention and treatment of bleeding episodes in PUPs.

ELIGIBILITY:
Key Inclusion Criteria:

* Weight >=3.5 kilogram at the time of informed consent.
* Severe hemophilia B was defined as less than or equal to (<=)2 International Units per deciliter (IU/dL) (<=2 percent [%]) endogenous FIX documented in the medical record or as tested during the Screening Period.

Key Exclusion Criteria:

* History of positive inhibitor testing. A prior history of inhibitors was defined based on a participant's historical positive inhibitor test using the local laboratory Bethesda value for a positive inhibitor test (that is equal to or above lower limit of detection).
* History of hypersensitivity reactions associated with any rFIXFc administration.
* Exposure to blood components or injection with a coagulation factor IX (FIX) concentrate (including plasma derived) other than rFIXFc.
* Injection with commercially available rFIXFc more than 28 days prior to Screening.
* More than 3 injections of commercially available rFIXFc prior to confirmation of eligibility.
* Other coagulation disorders in addition to hemophilia B.
* Any concurrent clinically significant major disease that, in the opinion of the Investigator, would have made the participant unsuitable for enrollment (example HIV infection with cluster of differentiation 4 (CD4) lymphocyte count less than (<)200 cells/microliter (mcL) or a viral load greater than (>)200 particles/mcL, or any other known congenital or acquired immunodeficiency).
* Current systemic treatment with chemotherapy and/or other immunosuppressant drugs. Use of steroids for treatment of asthma or management of acute allergic episodes or otherwise life-threatening episodes was allowed. Treatment in these circumstances should not have exceeded a 14-day duration.
* Participation within the past 30 days in any other clinical study involving investigational treatment.
* Current enrollment in any other clinical study involving investigational treatment.
* Inability to comply with study requirements.
* Other unspecified reasons that, in the opinion of the Investigator or Bioverativ, would have made the participant unsuitable for enrollment.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Max Age: 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (11):
  - Research Site, Sacramento, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, East Lansing, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
- Research Site, Westmead, New South Wales, Australia
- Research Site, Aarhus, Denmark
- France (2):
  - Hopital Cardiologique - CHU Lille, Lille, Nord
  - Research Site, Lyon, Rhone
- Research Site, Dublin, Ireland
- Italy (4):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Roma
- Research Site, Utrecht, Netherlands
- Research Site, Auckland, New Zealand
- Research Site, Warsaw, Poland
- Research Site, Malmo, Sweden
- United Kingdom (3):
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, Whitechapel, London
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Nolan B, Recht M, Rendo P, Falk A, Foster M, Casiano S, Rauch A, Shapiro A. Prophylaxis with recombinant factor IX Fc fusion protein reduces the risk of bleeding and delays time to first spontaneous bleed event in previously untreated patients with haemophilia B: A post hoc analysis of the PUPs B-LONG study. Eur J Haematol. 2024 Oct;113(4):485-492. doi: 10.1111/ejh.14252. Epub 2024 Jun 25. PMID 38922990
- [Derived] Nolan B, Klukowska A, Shapiro A, Rauch A, Recht M, Ragni M, Curtin J, Gunawardena S, Mukhopadhyay S, Jayawardene D, Winding B, Fischer K, Liesner R. Final results of the PUPs B-LONG study: evaluating safety and efficacy of rFIXFc in previously untreated patients with hemophilia B. Blood Adv. 2021 Jul 13;5(13):2732-2739. doi: 10.1182/bloodadvances.2020004085. PMID 34242387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 active centers in 11 countries. Participants were screened between 13-Nov-2014 to 23-Jul-2018.
Pre-assignment Details: A total of 38 participants were screened. A total of 33 participants were enrolled, 22 participants began study participation on episodic treatment regimen and 11 participants began study participation on prophylactic treatment regimen.
Groups:
- Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc): Participants received rFIXFc intravenous (IV) injection as follows: Prophylactic treatment regimen: started with rFIXFc 50 International Units per kilogram (IU/kg) weekly until a participant reached at least 50 exposure days (ED=24-hour period in which greater than or equal to (>=1) injection/dose of rFIXFc was given) to rFIXFc, withdrawal from study or end of study. Adjustments to dose and dosing interval was based on incremental recovery, subsequent Factor IX levels, physical activity, bleeding pattern, in accordance with local standards of care for prophylactic regimen (PR). Treatment with episodic (on demand) regimen can be initiated before PR at investigators discretion. Episodic (On demand; optional): rFIXFc at individual doses based on participant's clinical condition, type and severity of bleeding event until PR.
Period: Overall Study
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Started | 33
Episodic Treatment Regimen | 22 (Participants were treated in more than one regimen and counted in all categories wherever applicable)
Prophylactic Treatment Regimen | 28 (17 participants among the 22 who started in episodic regimen, switched to the prophylactic regimen.)
Completed | 27
Not Completed | 6
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Eligibility Criteria not fulfilled | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Safety Analysis Set which included all participants who received at least 1 dose of study rFIXFc.
Groups:
- Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc): Participants received rFIXFc IV injection as follows: Prophylactic treatment regimen: started with rFIXFc 50 IU/kg weekly until a participant reached at least 50 exposure days (ED=24-hour period in which >=1 injection/dose of rFIXFc was given) to rFIXFc, withdrawal from study or end of study. Adjustments to dose and dosing interval was based on incremental recovery, subsequent Factor IX levels, physical activity, bleeding pattern, in accordance with local standards of care for prophylactic regimen (PR). Treatment with episodic (on demand) regimen can be initiated before PR at investigators discretion. Episodic (On demand; optional): rFIXFc at individual doses based on participant's clinical condition, type and severity of bleeding event until PR.
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 0.60 [0.08 to 2.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22
  Black or African-American | 1
  Asian | 1
  American Indian or Alaska Native | 0
  Native Hawaiian or other Pacific Islander | 0
  Unknown or Not reported | 5
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Inhibitor Development as Measured by the Nijmegen-Modified Bethesda Assay
Description: Development of an inhibitor was defined as an inhibitor test result of >= 0.60 Bethesda units per milliliter (BU/mL) that was confirmed by a second test result of >=0.60 BU/mL from a separate sample, drawn 2 to 4 weeks after the date when the original sample was drawn, with both tests performed by the central laboratory using Nijmegen-modified Bethesda assay.
Time Frame: Up to 3 years
Population: Analysis performed on Safety Analysis set which included all participants who had received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
percentage of participants | 3.03 [0.08 to 15.76]

2. Secondary Outcome: Annualized Number of Bleeding Episodes (Spontaneous and Traumatic) Per Participant (Annualized Bleeding Rate [ABR])
Description: ABR was annualized number of bleeding episodes during efficacy period (EP) per participant normalized to a 1-year interval of time. Bleeding episodes were classified as: spontaneous if parent/caregiver/participant records bleeding event when there is no known contributing factor such as definite trauma or antecedent strenuous activity; and traumatic when there is known reason for bleed. ABR=(Number of bleeding episodes during EP/total number of days during EP)*365.25. EP reflects the sum of all intervals of time during which participants were treated with rFIXFc per treatment regimens excluding surgical/rehabilitation periods and large injection intervals (greater than [>]28 days). Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis performed on Full Analysis Set (FAS) which included all enrolled participants with at least 1 dose of study treatment. Here, number analyzed signifies number of FAS participants who were analyzed in each treatment regimen.
Measure: Median (Full Range); unit: episodes per participant per year
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
episodes per participant per year
  Episodic regimen: number analyzed (Participants) | 22
  Episodic regimen | 0.21 [0.0 to 6.8]
  Prophylaxis regimen: number analyzed (Participants) | 28
  Prophylaxis regimen | 1.24 [0.0 to 5.4]

3. Secondary Outcome: Annualized Number of Spontaneous Joint Bleeding Episodes
Description: Bleeding episodes were classified as spontaneous if parent/caregiver/participant records a bleeding event when there is no known contributing factor such as a definite trauma or antecedent "strenuous" activity. Annualized spontaneous joint bleeding episodes=(Total number of spontaneous joint bleeding episodes during efficacy period (EP) divided by total number of days during EP)*365.25. EP reflects the sum of all intervals of time during which participants were treated with rFIXFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals (>28 days). Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis performed on FAS. Here, number analyzed signifies number of FAS participants who were analyzed in each treatment regimen.
Measure: Median (Full Range); unit: episodes per participant per year
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
episodes per participant per year
  Episodic regimen: number analyzed (Participants) | 22
  Episodic regimen | 0.00 [0.0 to 5.6]
  Prophylaxis regimen: number analyzed (Participants) | 28
  Prophylaxis regimen | 0.00 [0.0 to 2.6]

4. Secondary Outcome: Number of rFIXFc Injections With Excellent or Good, Moderate or None Treatment Response Assessed Using a 4-Point Scale
Description: Using e-diary, each participant's parent/caregiver rated treatment response to any bleeding episode (BE) at approximately 8 to 12 hours from time of injection and prior to additional doses of rFIXFc given for same BE using 4-point scale:- 1=Excellent: abrupt pain relief and/or improvement in signs of bleeding within approximately 8 hours after initial injection; 2=Good: definite pain relief and/or improvement in signs of bleeding within approx. 8 hours after injection, but possibly requiring more than 1 injection after 24-48 hours for complete resolution; 3=Moderate: Probable/slight beneficial effect within 8 hours after initial injection and requires more than 1 injection and 4=None: No improvement or condition worsens within approx. 8 hours after initial injection. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis performed on FAS. Analysis was based on all injections. Here, number analyzed signifies number of responses to injections reported for each treatment regimen.
Measure: Count of Units; unit: responses to injections
Units Other Than Participants: responses to injections
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
Number analyzed (responses to injections) | 154
responses to injections
  Episodic regimen: number analyzed (responses to injections) | 80
  Episodic regimen: Excellent or Good | 22
  Episodic regimen: Moderate | 0
  Episodic regimen: None | 0
  Episodic regimen: Response not provided | 58
  Prophylaxis regimen: number analyzed (responses to injections) | 74
  Prophylaxis regimen: Excellent or Good | 50
  Prophylaxis regimen: Moderate | 6
  Prophylaxis regimen: None | 1
  Prophylaxis regimen: Response not provided | 17

5. Secondary Outcome: Total Number of Exposure Days (EDs)
Description: An ED was defined as a 24-hour period in which a participant received one or more doses of rFIXFc injections, with the time of the first injection of rFIXFc defined as the start of the ED. Participant who did not have a particular injection type were counted as having zero injections for that type.
Time Frame: Up to 3 years
Population: Analysis performed on safety analysis set.
Measure: Median (Full Range); unit: days
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
days | 76.0 [1 to 137]

6. Secondary Outcome: Total Annualized rFIXFc Consumption Per Participant for the Prevention and Treatment of Bleeding Episodes
Description: Total annualized rFIXFc consumption (in IU/kg) was calculated for each participant as: Annualized consumption = (Total IU/kg of rFIXFc during efficacy period (EP) divided by total number of days during EP)*365.25. EP reflects the sum of all intervals of time during which participants were treated with rFIXFc according to the treatment regimens of the study excluding surgical/rehabilitation periods and large injection intervals (> 28 days). Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Median (Full Range); unit: IU per kilogram per participant per year
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
IU per kilogram per participant per year
  Episodic regimen: number analyzed (Participants) | 22
  Episodic regimen | 203.2 [0 to 5719]
  Prophylaxis regimen: number analyzed (Participants) | 28
  Prophylaxis regimen | 3175.0 [2544 to 13164]

7. Secondary Outcome: Number of Injections of rFIXFc Required to Resolve a Bleeding Episode
Description: Number of injections of rFIXFc required to resolve a bleeding episode during efficacy period (EP) were reported. EP reflects the sum of all intervals of time during which participants were treated with rFIXFc according to the treatment regimens of the study excluding surgical/rehabilitation periods and large injection intervals (>28 days). All injections given from the initial sign of a bleed, until the last date/time within the bleed window were counted. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis performed on FAS. Here, number analyzed signifies number of bleeding episodes reported for each treatment regimen.
Measure: Median (Full Range); unit: injections
Units Other Than Participants: Bleeding episodes
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
Number analyzed (Bleeding episodes) | 85
injections
  Episodic regimen: number analyzed (Participants) | 22
  Episodic regimen: number analyzed (Bleeding episodes) | 27
  Episodic regimen | 1.0 [1 to 31]
  Prophylaxis regimen: number analyzed (Participants) | 28
  Prophylaxis regimen: number analyzed (Bleeding episodes) | 58
  Prophylaxis regimen | 1.0 [1 to 4]

8. Secondary Outcome: Average Dose Per Injection of rFIXFc Required to Resolve a Bleeding Episode
Description: The average dose of rFIXFc per injection per bleeding episode was calculated as the average of all doses (IU/kg) administered to treat the bleeding episode during efficacy period (EP). EP begins with the first treatment regimen dose of rFIXFc and ends with the last dose (regardless of the reason for dosing). Surgery/rehabilitation periods are not included in the EP. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: as for outcome 7
Measure: Median (Full Range); unit: IU/kg
Units Other Than Participants: Bleeding episodes
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
Number analyzed (Bleeding episodes) | 85
IU/kg
  Episodic regimen: number analyzed (Participants) | 22
  Episodic regimen: number analyzed (Bleeding episodes) | 27
  Episodic regimen | 88.50 [41.7 to 178.6]
  Prophylaxis regimen: number analyzed (Participants) | 28
  Prophylaxis regimen: number analyzed (Bleeding episodes) | 58
  Prophylaxis regimen | 71.92 [23.3 to 181.8]

9. Secondary Outcome: Change From Baseline in rFIXFc Incremental Recovery (IR)
Description: Blood samples were taken at trough and Cmax (maximum concentration) for assessment of incremental recovery, measured by the one-stage clotting assay. IR (International Units per deciliter [IU/dL] per IU/kg) = (Cmax for FIX activity - Pre-dose FIX activity) (IU/dL)/ Actual dose (IU/kg), where Cmax is 30 minute FIX activity post-dose and FIX activity less than (<)0.5 IU/dL was set to 0 IU/dL for calculation of IR.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, and 144
Population: Analysis performed on FAS. Here number analyzed signifies number of FAS participants with available data for each visit.
Measure: Median (Inter-Quartile Range); unit: IU/dL per IU/kg
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
Number analyzed (Participants) | 33
IU/dL per IU/kg
  Change at Week 12: number analyzed (Participants) | 14
  Change at Week 12 | 0.0 [-0.08 to 0.12]
  Change at Week 24: number analyzed (Participants) | 15
  Change at Week 24 | 0.0 [-0.17 to 0.15]
  Change at Week 36: number analyzed (Participants) | 18
  Change at Week 36 | -0.0 [-0.18 to 0.11]
  Change at Week 48: number analyzed (Participants) | 20
  Change at Week 48 | -0.0 [-0.13 to 0.03]
  Change at Week 60: number analyzed (Participants) | 17
  Change at Week 60 | -0.1 [-0.1 to 0.03]
  Change at Week 72: number analyzed (Participants) | 12
  Change at Week 72 | -0.1 [-0.20 to 0.07]
  Change at Week 84: number analyzed (Participants) | 10
  Change at Week 84 | -0.1 [-0.23 to -0.04]
  Change at Week 96: number analyzed (Participants) | 7
  Change at Week 96 | -0.1 [-0.14 to 0.03]
  Change at Week 108: number analyzed (Participants) | 4
  Change at Week 108 | -0.1 [-0.36 to -0.01]
  Change at Week 120: number analyzed (Participants) | 1
  Change at Week 120 | -0.1 [-0.1 to -0.1]
  Change at Week 132: number analyzed (Participants) | 1
  Change at Week 132 | -0.1 [-0.1 to -0.1]
  Change at Week 144: number analyzed (Participants) | 1
  Change at Week 144 | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to end of the study (up to 3 years) regardless of seriousness or relationship to investigational product.
Description: Reported AE are treatment-emergent AE i.e. AE that was present prior to receiving first injection of rFIXFc and subsequently worsened in severity, or was not present prior to receiving first injection but subsequently appeared before last visit/follow-up call, whichever came later. Analysis performed on safety analysis set.
Arm/Group | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc)
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 23/33
Other Adverse Events (participants affected / at risk) | 27/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc) (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Factor ix inhibition (Blood and lymphatic system disorders) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infusion site pustule (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral rash (Infections and infestations) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (9)
Head injury (Injury, poisoning and procedural complications) | 3 (8)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Spinal cord haematoma (Nervous system disorders) | 1 (1)
Tongue biting (Nervous system disorders) | 1 (1)
Prepuce redundant (Reproductive system and breast disorders) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 9 (9)
Haematoma (Vascular disorders) | 1 (1)
Poor venous access (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor IX Fc Fusion Protein (rFIXFc) (N=33)
Middle ear effusion (Ear and labyrinth disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (9)
Teething (Gastrointestinal disorders) | 6 (15)
Vomiting (Gastrointestinal disorders) | 4 (8)
Pyrexia (General disorders) | 14 (33)
Bronchitis (Infections and infestations) | 2 (4)
Conjunctivitis (Infections and infestations) | 2 (2)
Croup infectious (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 4 (4)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 11 (22)
Otitis media (Infections and infestations) | 4 (8)
Pharyngitis (Infections and infestations) | 4 (5)
Rhinitis (Infections and infestations) | 3 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (12)
Varicella (Infections and infestations) | 4 (4)
Viral infection (Infections and infestations) | 4 (6)
Viral rash (Infections and infestations) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 7 (13)
Head injury (Injury, poisoning and procedural complications) | 5 (7)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
White blood cell count increased (Investigations) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 3 (4)
Irritability (Psychiatric disorders) | 2 (2)
Balanoposthitis (Reproductive system and breast disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (18)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT02234310/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT02234310/SAP_001.pdf